CLINICAL TRIAL: NCT04335812
Title: Internet-based Cognitive Behavioral Therapy for Tinnitus Sufferers: Comparing the Full CBT Program With Relaxation Only Program
Brief Title: Internet-based Cognitive Behavioral Therapy for Tinnitus Sufferers
Acronym: ICBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lamar University (Other)
Responsible Party: Principal Investigator, Vinaya Manchaiah, Jo Mayo Endowed Professor, Lamar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-FY20-200-1
Record Dates: First submitted 2020-04-03; First posted 2020-04-06 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- R-ICBT (Experimental): The intervention offered is a guided relaxation-based CBT offered via the Internet. The intervention is similar to a self-help program, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is a 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice the techniques learned. The modules provided will focus on applied relaxation only.
  Interventions: Behavioral: Internet-based Cognitive Behavior Therapy
- F-ICBT (Active Comparator): The intervention offered is a guided Internet-based CBT intervention. The intervention is similar to a self-help program, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is a 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice the techniques learned. The modules are a mixture of applied relaxation, Cognitive Behavioral Therapy and advice addressing common problems
  Interventions: Behavioral: Internet-based Cognitive Behavior Therapy

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavior Therapy — The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned.
  Other Names: ICBT

SUMMARY:
Nearly 50 million people in the U.S. experience tinnitus, of which about 20 million people have burdensome chronic tinnitus. Tinnitus can be very debilitating as many aspects of daily life can be affected, such as sleep, mood, and concentration. Currently, there is no cure for tinnitus. Pharmacological or sound-therapy based interventions are sometimes provided but may be of limited value to certain individuals. Research suggests that Cognitive Behavior Therapy (CBT) based approaches have the most evidence of effectiveness in the management of tinnitus. However, CBT is rarely offered to tinnitus sufferers in the U.S. (less than 1%), partly because of lack of trained professionals who can deliver CBT. To improve access to CBT for tinnitus, an online CBT program has been developed. The purpose of this study is to evaluate if the full CBT administered via the Internet results in better outcomes when compared to relaxation only CBT administered via the Internet for adults with tinnitus in the United States.

DETAILED DESCRIPTION:
Objective: To examine the difference in outcomes of relaxation-based Internet-based cognitive behavioral therapy (R-ICBT) versus full version of Internet-based cognitive behavioral therapy (F-ICBT) for tinnitus sufferers.

Hypothesis: It is hypothesized that F-ICBT (experimental group) is superior when compared to R-ICBT (control group) in reducing the tinnitus-related distress, decreasing sleep disturbance, decreasing anxiety and depression, and improving health-related quality of life. The investigators also hypothesize that these results will be stable in both short- and long-term post-intervention.

Design: A two-armed Randomized Control Trial (RCT), with a one-year follow-up design will be used to evaluate the efficacy of F-ICBT and R-ICBT on tinnitus distress.

Setting: This will be an Internet-based study for adults with tinnitus living in the USA.

Participants: Eligible participants will include adults with tinnitus for a minimum period of 3 months with internet access and no major medical or psychiatric conditions. 100 participants will be recruited for each group and will be randomly assigned using a computer-generated randomization schedule by an independent research assistant after being pre-stratified for tinnitus severity and depression severity.

Intervention: The intervention offered to experimental group is a guided CTB-based internet intervention (ICBT), providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned. The experimental group will be given the full ICBT program with all the components (22 chapters), whereas the control group will get only the relaxation-based exercises (8 chapters) of the ICBT program.

Outcome measures: The main outcome measure is the Tinnitus Functional Index (TFI). Secondary outcome measures are the Tinnitus and Hearing Survey (THS), Tinnitus Cognition Questionnaire (TCQ), Patient Health Questionnaire (PHQ-9), Generalized Anxiety Disorder (GAD-7), Insomnia Severity Index (ISI), and EuroQol EQ-5D-5L VAS.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years and older living in the USA;
2. the ability to read and type in English;
3. no barriers to using a computer (e.g. no significant fine motor control or visual problems);
4. Internet and e-mail access and the ability to use it;
5. commitment to completing the program;
6. completion of the online screening and outcome questionnaires;
7. agree to participate in either group and be randomized to one of these groups;
8. understand and work towards the end goal of reducing the impact and distress of tinnitus, although the strength of the tinnitus may remain the same;
9. be available for 12 months after starting the study to complete a 1-year follow-up questionnaire; and
10. experience bothersome tinnitus for a minimum period of 3 months;

Exclusion Criteria:

1. reporting any major medical or psychiatric conditions;
2. reporting pulsatile, objective or unilateral tinnitus, which has not been investigated medically;
3. tinnitus as a consequence of a medical disorder, still under investigation; and
4. undergoing any other tinnitus therapy while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinaya Manchaiah, PhD, Principal Investigator — Lamar University
Locations (1):
- Lamar University, Beaumont, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are openly available in Figshare at https://doi.org/10.6084/m9.figshare.13679179
Supporting Information: Study Protocol, SAP
Time Frame: Available now
Access Criteria: Data are openly available
URL: https://doi.org/10.6084/m9.figshare.13679179

REFERENCES:
- [Result] Beukes EW, Andersson G, Fagelson MA, Manchaiah V. Dismantling internet-based cognitive behavioral therapy for tinnitus. The contribution of applied relaxation: A randomized controlled trial. Internet Interv. 2021 May 12;25:100402. doi: 10.1016/j.invent.2021.100402. eCollection 2021 Sep. PMID 34040997
- See also: Study website — http://www.tacklingtinnitus.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 135 participants completed the informed consent 9 participants were excluded (5 outside the country and 4 were no longer interested) 126 participants were included in the study
Period: Overall Study
Arm/Group | R-ICBT | F-ICBT
Started | 63 | 63
Completed | 28 | 30
Not Completed | 35 | 33
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 12 | 12
Not completed — Did not engage in the intervention | 22 | 18

BASELINE CHARACTERISTICS:
Groups:
- R-CBT: The intervention offered is a guided relaxation-based CBT offered via the Internet. The intervention is similar to a self-help program, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is a 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice the techniques learned. The modules provided will focus on applied relaxation only.
  Internet-based Cognitive Behavior Therapy: The intervention offered is a CTB-based internet intervention, providing an opportunity to learn about new ways of coping with tinnitus during everyday life. It is 8-week long e-learning intervention, with new modules introduced weekly and assignments are given to practice techniques learned.
- Total: Total of all reporting groups
Arm/Group | R-CBT | F-ICBT | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 55 (13) | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 37 | 62
  Male | 38 | 26 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 59 | 59 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 3 | 5
  White | 58 | 56 | 114
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 126
Tinnitus Functional Index (TFI) [Mean (Standard Deviation); unit: score on a scale] | 50.52 (26.65) | 48.70 (25.51) | 49.61 (26)

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Functional Index (TFI); Measure of Tinnitus Distress
Description: Tinnitus Functional Index (TFI) is a 25-item questionnaire that evaluates the severity of tinnitus distress. Total possible score ranges from 0-to-100 with higher scores suggesting more severe tinnitus distress (i.e., worse outcome). Scores >25 indicate tinnitus is a significant problem requiring tinnitus intervention.
Time Frame: T0: Baseline, T1: Post-intervention 1 (after both group complete initial intervention), T2: Post-intervention 2 (after R-ICBT group complete Full ICBT), T3: 2-months post-intervention
Population: 63 participants started the trial in both the R-ICBT (applied relaxation) and F-ICBT (full ICBT) groups 28 participants from the R-ICBT and 30 from the ICBT completed the post-intervention measure 29 participants from the R-ICBT and 30 from the ICBT completed the post-intervention measure after both groups completed full ICBT 23 participants from the R-ICBTgroup and 19 from the ICBT group completed the 2-month post-intervention measure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 48.7 (25.51) | 50.52 (26.65)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 32.13 (21.38) | 28.95 (20.75)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 30.66 (23.45) | 28.95 (20.75)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 23.81 (9.87) | 27.16 (20.78)

2. Secondary Outcome: Tinnitus Cognition Questionnaire (TCQ); Measure of Tinnitus Cognition
Description: Tinnitus Cognition Questionnaire (TCQ) is a 26-item questionnaire that assesses positive and negative cognitions associated with tinnitus. The first 13 items refer to negative thoughts and the second 13 items refer to positive thoughts. Responses are marked on a five-point Likert scale (0 to 4). The negative items (1-13) are scored 0-4, whereas the positive items (14-26) are reverse-scored: 4-0. The scoring procedure involves the simple addition of the number circled by the respondent for items 1-13 and the addition of reverse-scored items 14-26. The total score of the TCQ has a potential range from 0 to 104. A high score represents a greater tendency to engage in negative cognitions (i.e., worse outcome) in response to tinnitus and low engagement in positive cognitions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 44.67 (20.43) | 42.52 (18.58)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 30.96 (20.03) | 27.26 (20.17)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 28.93 (17.81) | 27.26 (20.17)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 25.30 (15.84) | 23.07 (17.54)

3. Secondary Outcome: Patient Health Questionnaire (PHQ-9); Measure of Depression
Description: Patient Health Questionnaire (PHQ-9) is a 9-item questionnaire that assesses depression severity. Responses are marked on a four-point Likert scale (0 to 3). The total score can range from 0 to 27 with higher scores indicating more severe depression (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 9.17 (7.12) | 9.10 (7.14)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 4.96 (5.07) | 4.32 (3.95)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 5.04 (5.7) | 4.32 (3.95)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 3.35 (4.17) | 4.12 (4.4)

4. Secondary Outcome: Generalized Anxiety Disorder (GAD-7); Measure of Anxiety
Description: Generalized Anxiety Disorder (GAD-7) is a 7-item questionnaire that assesses the severity of anxiety. Responses are marked on a four-point Likert scale (0 to 3). The total score can range from 0 to 21 with higher scores indicating more severe anxiety (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 7.75 (6.77) | 9.19 (6.39)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 5.21 (5.62) | 4.48 (4.17)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 4.86 (5.84) | 4.48 (4.17)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 3.70 (3.88) | 4.68 (4.75)

5. Secondary Outcome: Insomnia Severity Index (ISI); Measure of Insomnia
Description: Insomnia Severity Index (ISI) is a 7-item questionnaire that evaluates insomnia. Responses are marked on a five-point Likert scale (0 to 4). The total score can range from 0 to 28 with higher scores indicating more severe insomnia (i.w., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 11.90 (7.45) | 12.25 (7.7)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 8.93 (6.5) | 7.46 (5.8)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 8.43 (5.93) | 7.46 (5.8)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 7.13 (5) | 6.33 (6.08)

6. Secondary Outcome: EuroQol EQ-5D-5L VAS; Measure of Health-related Quality of Life
Description: EQ-5D-5L VAS is a single-item questionnaire that evaluates the health-related quality of life. Responses are marked on a 0-100 scale with higher scores indicating higher health-related quality o life (i.e., better outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 72.59 (17) | 75.43 (15.92)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 79.71 (12.14) | 78.15 (17.51)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 76.43 (15.79) | 78.15 (17.51)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 78.22 (11.29) | 85.87 (6.91)

7. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Tinnitus Sub-scale; Measure of Tinnitus Problem
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problem and ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). The total THS score can range from 0 to 40. However, the scores for this specific sub-scale can range from 0 to 16 with higher scores indicating more tinnitus problem (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 5.79 (4.55) | 6.29 (5.70)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 3.21 (3.32) | 2.85 (2.66)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 3.36 (3.68) | 2.85 (2.66)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 2.78 (3.19) | 2.07 (2.12)

8. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Hearing Sub-scale; Measure of Hearing Problem
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problem and ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). The total THS score can range from 0 to 40. However, the scores for this specific sub-scale can range from 0 to 16 with higher scores indicating more hearing problem (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 6.19 (4.84) | 5.94 (5.06)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 3.75 (3.7) | 4.59 (4.01)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | 4.71 (4.32) | 4.59 (4.01)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 4.65 (3.59) | 3.13 (2.36)

9. Secondary Outcome: Tinnitus and Hearing Survey (THS) - Sound Tolerance Sub-scale; Measure of Sound Tolerance
Description: Tinnitus and Hearing Survey (THS) is a 10-item questionnaire that helps in determining how much of a patient's complaint about tinnitus is due to a hearing problem and how much is due specifically to the tinnitus. THS has three sections/subscales (A, B, and C). Section A consists of four items that address common tinnitus problems. Section B contains four items that address hearing. Section C, which includes two items, which focus on sound tolerance problem and ability to participate in group therapy. Responses for each item can range from 0 (not a problem) to 4 (very big problem). The total THS score can range from 0 to 40. However, the scores for this specific sub-scale can range from 0 to 8 with higher scores indicating more sound tolerance problem (i.e., worse outcome).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | R-ICBT | F-ICBT
Number analyzed (Participants) | 63 | 63
score on a scale
  T0: Baseline | 1.17 (1.4) | 1.22 (1.3)
  T1: Post-intervention 1: number analyzed (Participants) | 28 | 30
  T1: Post-intervention 1 | 1.0 (1.39) | 0.67 (1.07)
  T2: Post-intervention 2 (both completed full ICBT): number analyzed (Participants) | 29 | 30
  T2: Post-intervention 2 (both completed full ICBT) | .96 (1.3) | .67 (1.07)
  T3: 2-month post-intervention: number analyzed (Participants) | 23 | 19
  T3: 2-month post-intervention | 0.91 (1.08) | 0.47 (0.74)

ADVERSE EVENTS:
Time Frame: T0: Baseline, T1: Post-intervention 1 (after both group complete initial intervention), T2: Post-intervention 2 (after R-ICBT group complete Full ICBT), T3: 2-months post-intervention
Description: Our definition of adverse events is the same as clinical trials.gov.
Arm/Group | R-ICBT | F-ICBT
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

LIMITATIONS AND CAVEATS:
The study was done during the height of the COVID-19 pandemic, during a time where day-to-day living was disrupted for most people. This may have been one of the key reasons for poor engagement with the intervention and poor compliance with the completion of outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04335812/Prot_SAP_000.pdf